CLINICAL TRIAL: NCT02096042
Title: A Phase I/II Study of Weekly Schedule Of Brentuximab Vedotin Alone and In Combination With 5-Azacytidine In Cluster of Differentiation Antigen (CD30)-Positive Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Phase I/II - Brentuximab/5-Azacytidine in Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0706; NCI-2014-01114 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia; AML; CD30-Positive; Relapsed; Refractory; Brentuximab Vedotin; SGN-35; Adcetris; 5-Azacytidine; Azacytidine; Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Recurrence | interventions — Brentuximab Vedotin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brentuximab Vedotin (Experimental): Pilot Phase: Starting dose of Brentuximab Vedotin 1.2 mg/kg intravenous (IV) infusion over approximately 30 minutes on days 1, 8, and 15 of each 28-day cycle (+/- 3 days).
  Interventions: Drug: Brentuximab Vedotin
- Brentuximab Vedotin + 5-Azacytidine (Experimental): Phase I Dose-Escalation Phase: Starting dose of Brentuximab Vedotin 1.0 mg/kg IV (starting dose level 1), or one-dose level lower than the established MTD if the pilot portion of the study establishes a lower MTD, infusion over approximately 30 minutes on days 1, 8, and 15 of each 28-day cycle. All patients receive 5-azacytidine at 75 mg/m2/day by vein or subcutaneously on days 1-7 every 28 days.
  Phase II Dose-Expansion Phase: Patients receive Brentuximab Vedotin at MTD from dose-escalation phase by vein on Days 1, 8, and 15 of each 28-day cycle. Patients receive 5-Azacytidine at 75 mg/m2/day by vein or subcutaneously on days 1-7 every 28 days. Patients can receive up to a total of 12 cycles of treatment (weekly + monthly combined).
  Interventions: Drug: Brentuximab Vedotin; Drug: 5-Azacytidine

INTERVENTIONS:
Drug: Brentuximab Vedotin — Pilot Phase: Starting dose of Brentuximab Vedotin 1.2 mg/kg intravenous (IV) infusion over approximately 30 minutes on days 1, 8, and 15 of each 28-day cycle.
  Phase I Dose-Escalation Phase: Starting dose of Brentuximab Vedotin 1.0 mg/kg IV (starting dose level 1), or one-dose level lower than the established MTD if the pilot portion of the study establishes a lower MTD, infusion over approximately 30 minutes on days 1, 8, and 15 of each 28-day cycle.
  Phase II Dose-Expansion Phase: Patients receive Brentuximab Vedotin at MTD from dose-escalation phase by vein on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: SGN-35; Adcetris
Drug: 5-Azacytidine — Phase I Dose-Escalation Phase and Phase II Dose-Expansion Phase: 5-Azacytidine at 75 mg/m2/day by vein or subcutaneously on days 1-7 every 28 days.
  Other Names: Azacytidine; Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Brentuximab Vedotin + 5-Azacytidine

SUMMARY:
This clinical research study is made up of 3 phases: a Pilot Phase, Phase 1, and Phase 2.

The goal of the Pilot Phase is to learn how safe it is to give the study drug brentuximab vedotin to patients with AML. The goal of Phase 1 is to learn more about the safety of the combination of brentuximab vedotin with azacytidine. The goal of Phase 2 is to learn if the combination of brentuximab vedotin and azacytidine can help to control AML.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of 3-6 participants will be enrolled in the Pilot Phase, up to 3 groups of 3-6 participants will be enrolled in Phase I of the study, and up to 25 participants will be enrolled in Phase II.

If you are enrolled in the Pilot Phase, the dose of brentuximab vedotin you receive will depend on when you joined this study. The first group of participants will receive the highest dose level of brentuximab vedotin. If intolerable side effects are seen, up to 2 more groups will be enrolled and will receive a lower dose of brentuximab vedotin than the group before it. If intolerable side effects are not seen, the next phase of the study will begin.

If you are enrolled in Phase I, the dose of brentuximab vedotin you receive will depend on when you joined this study. The first group of participants will receive a lower dose level of brentuximab vedotin than the highest one that was tolerated in the Pilot Phase, and will also receive azacitidine. If intolerable side effects are seen, up to 2 more groups will be enrolled and will receive a lower dose of brentuximab vedotin than the group before it. If intolerable side effects are not seen, the next phase of the study will begin.

If you are enrolled in Phase 2, you will receive brentuximab vedotin at the highest dose that was tolerated in Phase 1.

All participants in Phases 1 and 2 will receive the same dose level of azacytidine.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive brentuximab vedotin by vein over 30 minutes on Days 1, 8, and 15 of each 28-day study cycle. If the disease appears to get better, or after cycle 4, the dose and schedule of brentuximab vedotin may be changed to monthly rather than weekly doses.

If you are in Phase 1 or Phase 2, you will also receive azacytidine by vein or as an injection under the skin on Days 1-7 of each cycle.

You may be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

On Day 1 of each cycle:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* You will have an EKG.
* Every 3 Cycles (Cycles 3, 6, 9, and so on), if you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

On Days 8 and 22 of Cycle 1, blood (about 2-3 tablespoons) will be drawn for routine tests.

On Day 15 of Cycle 1:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.

On Day 28 of Cycle 1, then Day 1 of every 2 cycles after that (Cycles 3, 5, 7, and so on), you will have a bone marrow biopsy and/or aspirate to check the status of the disease. After any point that the disease appears to get better, this will be done every 3-4 cycles, or whenever your doctor thinks it is needed.

Length of Treatment:

You may receive the study drug for up to 12 cycles. You will no longer be able to receive the study drug(s) if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the end-of-study visit.

End-of-Study Visit:

About 28 days after your last dose of study drug, you will have an end-of-study visit:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* You will have an EKG to check your heart function.
* You may have a bone marrow biopsy and/or aspirate to check the status of the disease.
* If you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

If the End-of-Study Visit occurs within 21 days of your last dose, you will be called by a member of the study team about 30-37 days after your last dose of study drug. You will be asked how you are feeling and about any side effects you may be having. This call will last about 5 minutes.

This is an investigational study. Brentuximab vedotin is FDA approved and commercially available for the treatment of certain types of lymphoma after previous treatments have failed. Its use in combination with azacitidine is investigational. Azacytidine is FDA approved and commercially available for the treatment of myelodysplastic syndrome (MDS) and chronic myelomonocytic leukemia (CMML).

The study doctor can explain how the study drug(s) are designed to work.

Up to 61 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed AML, other than acute promyelocytic leukemia, as defined by the 2008 World Health Organization (WHO) criteria that is relapsed or refractory to standard chemotherapy. Note: Newly-diagnosed AML patients who are 60 years or older and are not candidates for or have refused standard chemotherapy are also eligible for this trial.
2. AML blasts must express CD30 (>/=10% expression as assessed by flow-cytometry or 2+ expression by immunohistochemistry) (whenever possible CD30 expression will be assessed by both methods)
3. Age 18 years or older
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of </=3
5. The following baseline laboratory data: Serum bilirubin </=1.5 x upper limit of normal (ULN) or </= 3 x ULN for patients with Gilbert's disease; Serum creatinine </=1.5 x ULN AND creatinine clearance >30 ml/min; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </=3 x ULN
6. Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (beta-hCG) pregnancy test result within 14 days prior to the first dose of brentuximab vedotin and must agree to use an effective contraception method during the study and for 30 days following the last dose of study drug. Females of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy.
7. Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
8. Patients or their legally authorized representative must provide written informed consent.

Exclusion Criteria:

1. History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses).
2. Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association Class III-IV within 6 months prior to their first dose of brentuximab vedotin
3. Evidence of active cerebral/meningeal disease. Patients may have history of central nervous system (CNS) leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of registration.
4. Previous treatment with any anti-CD30 directed therapy
5. Patients with previous allogeneic stem cell transplant (SCT) if they meet either of the following criteria: <100 days from allogeneic SCT, Acute or chronic graft-versus-host disease (GvHD), or Receiving immunosuppressive therapy as treatment for or prophylaxis against GvHD within the last 7 days
6. Patients with uncontrolled active infections (viral, bacterial, and fungal) are not eligible.
7. Known to be positive for hepatitis B by surface antigen expression
8. Known to have active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months)
9. Preexisting grade >/=2 peripheral neuropathy
10. Patients with uncontrolled diabetes mellitus
11. Current therapy with other systemic anti-neoplastic or anti-neoplastic investigational agents.
12. Chemotherapy (except hydroxyurea or emergent use of single-agent cytarabine for cytoreduction), radiotherapy, biologics, and/or other treatment with immunotherapy that is not completed 2 weeks prior to first dose of study drug, unless progressive disease is documented. NOTE: Hydroxyurea will be allowed during the first cycle of treatment
13. Females who are pregnant or lactating
14. Known hypersensitivity to any excipient contained in the drug formulation of brentuximab vedotin
15. History of progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 24, 2014 to July 08, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study was terminated early due to low enrollment.
Groups:
- Brentuximab Vedotin + 5-Azacytidine: Phase I Dose-Escalation Phase: Starting dose of Brentuximab Vedotin 1.0 mg/kg IV (starting dose level 1), or one-dose level lower than the established MTD if the pilot portion of the study establishes a lower MTD, infusion over approximately 30 minutes on days 1, 8, and 15 of each 28-day cycle. 5-azacytidine at 75 mg/m2/day IV or subcutaneously on days 1-7 every 28 days.
- MTD Brentuximab Vedotin + 5-Azacytidine: Phase II Dose-Expansion Phase: Brentuximab Vedotin at MTD from dose-escalation phase IV on Days 1, 8, and 15 of each 28-day cycle. 5-Azacytidine at 75 mg/m2/day IV or subcutaneously on days 1-7 every 28 days.Up to 12 cycles of treatment (weekly + monthly combined).
Period: Overall Study
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + 5-Azacytidine | MTD Brentuximab Vedotin + 5-Azacytidine
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Brentuximab Vedotin in Combination With 5-Azacytidine
Description: MTD defined as maximum dose at which <33% of patients experience a dose-limiting toxicity (DLT) during cycle 1.
Time Frame: After 1, 28 day cycle
Population: Study terminated early.
Arm/Group | Brentuximab Vedotin + 5-Azacytidine
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Response Rate
Description: Response defined as number of participants with complete response (CR), CR with incomplete platelet recovery (CRp), CR with insufficient hematological recovery (CRi) or partial remission (PR).
Time Frame: Response assessed after four 28-day cycles, up to 120 days
Population: Study was stopped with only one participant; no analysis done on outcome.
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + 5-Azacytidine | MTD Brentuximab Vedotin + 5-Azacytidine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection for first 28-day cycle.
Arm/Group | Brentuximab Vedotin
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin (N=1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes